CLINICAL TRIAL: NCT05398081
Title: Comparative Efficacy of Intravenous Cefuroxime and Ceftriaxone in Preventing Surgical Site Infection After Neurosurgical Procedures
Brief Title: Cefuroxime vs Ceftriaxone for SSI Prevention in Neurosurgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Promise Tamunoipiriala Jaja (Other)
Responsible Party: Sponsor-Investigator, Dr. Promise Tamunoipiriala Jaja, Doctor, University College Hospital, Ibadan
Organization: University College Hospital, Ibadan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UI/EC/21/0099
Record Dates: First submitted 2021-12-26; First posted 2022-05-31 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Surgical Site Infection; Antibiotics Prophylaxis
Keywords: Surgical site infection; Antibiotics prophylaxis; Cefuroxime; Ceftriaxone; Craniotomy; Laminectomy
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefuroxime; cefuroxime axetil; Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cefuroxime (Experimental): Cefuroxime (Zinnat®) will be used as prophylactic antibiotic in this arm
  Interventions: Drug: Cefuroxime (Zinnat®)
- Ceftriaxone (Active Comparator): Ceftriaxone (Rocephin®) will be used as prophylactic antibiotic in this arm
  Interventions: Drug: Ceftriaxone (Rocephin®)

INTERVENTIONS:
Drug: Cefuroxime (Zinnat®) — Antibiotic for prophylaxis against surgical site infection following craniotomy and laminectomy Here, Cefuroxime (Zinnat®), a second generation cephalosporin will be used
  Arms: Cefuroxime
Drug: Ceftriaxone (Rocephin®) — Antibiotic for prophylaxis against surgical site infection following craniotomy and laminectomy Here, Ceftriaxone (Rocephin®) a third generation cephalosporin will be used
  Arms: Ceftriaxone

SUMMARY:
BACKGROUND: Surgical site infection (SSI) is potentially catastrophic in neurosurgical procedures, causing poor in-hospital outcomes in more than half of those affected and significantly increased length of hospital stay. The appropriate and timely use of prophylactic antibiotics is found to reduce the prevalence of SSIs. At present, several regimen of antimicrobial agents are used in neurosurgical procedures since the choice of appropriate antibiotic agent is not fully established. Cephalosporins are among the frequently used antibiotics for prophylaxis in neurosurgical procedures, with studies comparing first and second generation Cephalosporins to third generation in neurosurgical prophylaxis, showing no superiority of the latter over the former. Clearly, comparing Cefuroxime (a second generation Cephalosporin) to Ceftriaxone (a third generation Cephalosporin) in neurosurgical procedures will provide more knowledge on the efficacy of Cefuroxime as antibiotics prophylaxis.

OBJECTIVE: The study aimed to determine the comparative efficacy of cefuroxime versus ceftriaxone in the prevention of surgical site infection after neurosurgical procedures at the University College Hospital Ibadan, Nigeria.

METHODS: The study will be a randomized controlled trial recruiting 92 participants. Participants would be patients undergoing neurosurgical procedures; they will be randomized to treatment arms (those receiving cefuroxime versus ceftriaxone for antibiotic prophylaxis). All the study articipants will be followed up for 30 days to assess for the development of surgical site infection.

DATA ANALYSIS: Data will be collated, computed and analyzed using the Statistical Product and Service Solutions (SPSS) Version 21. Demographics will be presented using summary statistics; mean +/- standard deviation and figures (e.g pie chart, histogram). Study outcomes will yield categorical and continuous variables which will be analyzed using chi-squared test and Z-test and/or T-test for hypothesis testing.

DETAILED DESCRIPTION:
BACKGROUND Surgical Site Infection (SSI) is the most common health care-associated infection in hospitalized patients, accounting for 31% of all infections globally.

The prevalence of SSI is determined by the antibiotics prophylaxis, the duration of postoperative monitoring, the institution and the type of surgical procedures. It ranges between 1% and 17% in most surgical specialties. In the Sub-Saharan Africa, the prevalence of SSI following neurosurgical procedures when two different third-generation cephalosporins were used as antibiotic prophylaxis in the same institution were 6.9% and 15% respectively. It is indeed catastrophic, causing poor in-hospital outcomes in upwards of half of those affected and significantly increased their length of hospital stay. SSI following craniotomy costs an average of ₤9,283 above the initial cost of treatment to manage, in addition to the prolonged disablement and reduced functioning of the patient.

Appropriate and timely use of prophylactic antibiotics reduced the prevalence of SSIs from 8.8% to 4.6%. At present, several regimen of antimicrobial agents are used in neurosurgical procedures in the absence of a 'choice' antibiotic agent. The choice, ideal antibiotics should have an appropriate antimicrobial spectrum and favourable pharmacokinetics.

Cephalosporin is among the frequently used antibiotics for prophylaxis in neurosurgical procedures due to its wide spectrum of their effectiveness, good tissue penetration, and the low toxicity of its first and second generation agents. They are bactericidal agents, with a beta-lactam ring structure that determines their antibacterial activity and a six-member dihydrothiazine ring which is responsible for their ability to resist inactivation by certain bacterial enzymes. They have different antibacterial activity based on substitutions at position 7 of the Cephalosporin nucleus. Following penetration of the bacterial cell surface, they attach to bacterial penicillin-binding proteins - proteins thay catalyze critical cell-wall synthesis and division reactions; thus interrupting of bacterial cell-wall synthesis and division.

The first and second-generation Cephalosporins also have the pharmacological advantage that in case of postoperative infection the third and other newer generation Cephalosporin can be given with only a slight chance of developing early resistance.Third generation Cephalosporins, due to their better coverage of gram-negative bacteria compared to the first and second generation agents, have somewhat been put forward since some noticeable change in spectrum toward more gram-negative bacteria has been observed in the microbiological profiles of some series on SSI. Mainly gram-positive cocci; (especially S.aureus and S.epidermidis) are associated with SSI in neurosurgery.

The widespread use of the third generation Cephalosporin has been associated with an increase in Extended Spectrum β-Lactamase(ESBL)- mediated resistance amongst Gram-negative pathogens, as well as antibiotic-associated diarrhea due to Clostridium-difficile and Methicillin Resistant Staphylococcus Aureus(MRSA) and Enterococci. Therefore, there is the need to restrict the use of third generation Cephalosporins for perioperative prophylaxis in neurosurgery.

There are studies which have compared first and second generation Cephalosporins to third generation in neurosurgical prophylaxis, showing no any superiority of the latter over the former. Cefuroxime is a second-generation cephalosporin effective against Staphylococcus aureus, groups A and B streptococci, and S pneumonia. It has moderate activity against a limited number of aerobic Gram-negative bacilli: Escherichia coli, Klebsiella pneumoniae and Proteus mirabilis, while it is inactive against anaerobic bacteria.

STATEMENT OF PROBLEM The enhanced activities of third-generation cephalosporins and other novel beta-lactam antibiotics, such as Cefotaxime, Ceftriaxone, Ceftazidime, and Imipenem, are directed against multi-resistant aerobic gram-negative bacilli, which are exceptional causes of postoperative infection in neurosurgical patients. These drugs are therefore conceptually inappropriate for prophylaxis, but are the ones most commonly used, if not the sole agents of, surgical prophylaxis in most neurosurgical procedures in this environment. Clearly comparing Cefuroxime a second generation Cephalosporin to Ceftriaxone a third generation Cephalosporin in neurosurgical procedures in this environment will help resolve the question of whether the more microbiologically-sound use of lower-generation antimicrobial agent in surgical prophylaxis is safe, and if so, can help spare and preserve the higher-generation agent for more specific use and also, it will help to improve knowledge on the efficacy of Cefuroxime as antibiotics prophylaxis in this environment. It is therefore hypothesized that second-generation cephalosporins like Cefuroxime would be no less effectual than the currently preferred third-generation agents (Ceftriaxone, Ceftazidime) in operative neurosurgical prophylaxis.

GENERAL OBJECTIVE:

The aim of this study is to compare the effectiveness of two perioperative prophylactic antibiotic regimens Cefuroxime (second generation Cephalosporin) and Ceftriaxone (third generation Cephalosporin) in the prevention of surgical site infection after neurosurgical procedures in the University College Hospital Ibadan, Nigeria.

SPECIFIC OBJECTIVES:

To determine the incidence of surgical site infection after clean and clean-contaminated neurosurgical procedures at the University College Hospital, Ibadan To determine the bacterial spectrum with the use of cefuroxime and ceftriaxone for antibiotic prophylactic regimen for neurosurgical procedures.

To determine the cost of antibiotic prophylaxis regimens in neurosurgical procedure in each sub-group

NULL HYPOTHESIS Cefuroxime would be less effectual than the currently preferred third-generation cephalosporin agents such as Ceftriaxone in neurosurgical prophylaxis.

ALTERNATE HYPOTHESIS Cefuroxime would be no less effectual than the currently preferred third generation cephalosporin agents such as Ceftriaxone and in neurosurgical prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for clean and clean-contaminated neurosurgical procedures that consent to participating in the study.

Exclusion Criteria:

* Patients with contaminated and dirty wounds e.g. grossly contaminated open depressed skull fracture, cranial endonasal surgeries and so on.
* Patients who has had systemic antibiotic therapy within 7 days before surgery.
* Patients with diabetes mellitus.
* Patients with implants (they will need longer follow up).
* Allergy to cephalosporins
* Infectious disease such as brain abscess, subdural empyema, osteitis and scalp infection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-06 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | Six weeks
  The presence or absence surgical site infection
Types and number of organism(s) causing surgical site infection | Six weeks
  The organisms isolated following culture of samples from an area of surgical site infection will be identified and a count will be made.

SECONDARY OUTCOMES:
Cost of care | Six weeks
  The cost of antibiotic prophylaxis in each sub-group will be determined in collaboration with the hospital pharmacy department.

CONTACTS AND LOCATIONS:
Overall Officials: Oghenekevwe E Okere, MBBS, Principal Investigator — University College Hospital, Ibadan; Amos O Adeleye, FWACS, FACS, Study Director — University College Hospital, Ibadan; Augustine A Adeolu, FWACS, Study Director — University College Hospital, Ibadan
Locations (1):
- University College Hospital, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant will be prepared and kept in data repositories
Supporting Information: Study Protocol, SAP, ICF
Time Frame: About the year following completion of the study
Access Criteria: Access will be granted following request for permissions